CLINICAL TRIAL: NCT05841784
Title: NYU HARP Telephone-Based Mindfulness Program
Brief Title: HARP Mindfulness Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-01609
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MBCT-T (Reference) (Active Comparator): Participants will receive Mindfulness-Based Cognitive Therapy delivered via Telephone (MBCT-T).
  Interventions: Behavioral: MBCT-T
- MBCT-T + Booster Mindfulness Sessions (Experimental): Participants will receive Mindfulness-Based Cognitive Therapy delivered via Telephone (MBCT-T), in addition to booster mindfulness sessions.
  Interventions: Behavioral: MBCT-T; Behavioral: Booster Mindfulness Sessions
- MBCT-T + Website Support (Experimental): Participants will receive Mindfulness-Based Cognitive Therapy delivered via Telephone (MBCT-T), in addition to website support.
  Interventions: Behavioral: MBCT-T; Behavioral: Website Support
- MBCT-T + Website Support + Booster Mindfulness Sessions (Experimental): Participants will receive Mindfulness-Based Cognitive Therapy delivered via Telephone (MBCT-T), in addition to both booster sessions and website support.
  Interventions: Behavioral: MBCT-T; Behavioral: Booster Mindfulness Sessions; Behavioral: Website Support

INTERVENTIONS:
Behavioral: MBCT-T — MBCT-T is an 8-week group-based program that combines training in mindfulness and cognitive-behavioral therapy to reduce psychological distress and negative emotions. Each weekly 1-hour session will consist of a check-in, discussion, teaching, mindfulness or cognitive behavioral practice or exercise, inquiry by the facilitator, and summary of the at-home practice.
Behavioral: Booster Mindfulness Sessions — Following the standard 8-week MBCT-T program, participants in certain arms will receive monthly MBCT-T booster sessions for 4 months of follow up. Each booster session will be 1 hour long. The sessions will include a concise review and summary of the main MBCT-T sessions.
  Arms: MBCT-T + Booster Mindfulness Sessions; MBCT-T + Website Support + Booster Mindfulness Sessions
Behavioral: Website Support — Participants in certain arms will receive continuous intervention support via the use of an online study website. The website will provide quick access to intervention materials and support to encourage participants to complete the at-home practice and apply the content of the MBCT-T program to real life situations.
  Arms: MBCT-T + Website Support; MBCT-T + Website Support + Booster Mindfulness Sessions

SUMMARY:
This study was designed using the Multiphase Optimization Strategy (MOST) framework to determine whether two supplemental components increase the efficacy of a mindfulness-based cognitive therapy program delivered via telephone (MBCT-T) for psychological distress. Specifically, this study will test mindfulness booster sessions to follow a standard 8-week MBCT-T intervention, as well as website support in patients with heart disease and/or heart disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting one of the following criteria:

  * Has a diagnosis of ischemic heart disease (ICD-10 codes I20 - I25) with no cardiac hospitalizations in the past 6 months
  * Has cardiovascular disease risk factors without meeting a diagnosis of ischemic heart disease or having a cardiovascular disease event (heart attack, stroke, heart failure, and/or unstable angina). Cardiovascular disease risk factors include hypertensive diseases (ICD-10 codes I10 - I11, I15 - I16), diabetes (E8 - E13), and/or hyperlipidemia (E78.0 - E78.5, E78.9)
* Patients meeting one or more of the following criteria at baseline:

  * Elevated stress (PSS-10 score ≥15)
  * Mild to moderate depressive symptoms (PHQ-9 score between 5-14)
  * Mild or greater anxiety (GAD-7 score ≥5)
* Willing to provide informed consent and comply with all aspects of the protocol
* Able to read and communicate in English

Exclusion Criteria:

* Active suicidal ideation
* History of, or current diagnosis of, psychosis
* Significant cognitive impairment (noted in the EHR or evident during screening)
* Significant hearing loss
* Current participation in another behavioral clinical trial
* Has received the MBCT-T intervention in a previous clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite Score of 3 Questionnaires: Perceived Stress Scale 10-item Version (PSS-10); Patient Health Questionnaire 9-Item Version (PHQ-9); and Generalized Anxiety Disorder Questionnaire 7-Item Version (GAD-7) at Baseline | Baseline
  Composite score of 3 questionnaires. The total composite score is the sum of scores from the questionnaires and ranges from 0 to 88; lower scores indicate greater overall health.
  PSS-10 measures perceived stress over the past month. Items rated on a 5-point scale ranging from 0 (never) to 4 (very often). Total scores range from 0-40; higher scores indicate greater levels of perceived stress.
  PHQ-9 assesses depressive symptoms in the past two weeks. Items rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms.
  GAD-7 measures anxiety symptoms in the past 2 weeks. Items rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with recommended cutoffs for mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Composite Score of 3 Questionnaires: PSS-10; PHQ-9; and GAD-7 at Post-Intervention | Month 2
  Composite score of 3 questionnaires. The total composite score is the sum of scores from the questionnaires and ranges from 0 to 88; lower scores indicate greater overall health.
  PSS-10 measures perceived stress over the past month. Items rated on a 5-point scale ranging from 0 (never) to 4 (very often). Total scores range from 0-40; higher scores indicate greater levels of perceived stress.
  PHQ-9 assesses depressive symptoms in the past two weeks. Items rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms.
  GAD-7 measures anxiety symptoms in the past 2 weeks. Items rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with recommended cutoffs for mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Composite Score of 3 Questionnaires: PSS-10; PHQ-9; and GAD-7 at Follow-Up | Month 6
  Composite score of 3 questionnaires. The total composite score is the sum of scores from the questionnaires and ranges from 0 to 88; lower scores indicate greater overall health.
  PSS-10 measures perceived stress over the past month. Items rated on a 5-point scale ranging from 0 (never) to 4 (very often). Total scores range from 0-40; higher scores indicate greater levels of perceived stress.
  PHQ-9 assesses depressive symptoms in the past two weeks. Items rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms.
  GAD-7 measures anxiety symptoms in the past 2 weeks. Items rated on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with recommended cutoffs for mild (5-9), moderate (10-14), and severe (15-21) anxiety.

SECONDARY OUTCOMES:
PSS-10 Score at Baseline | Baseline
  The PSS-10 is used to measure perceived stress over the past month. Items are rated on a 5-point scale ranging from 0 (never) to 4 (very often). Total scores range from 0-40; higher scores indicate greater levels of perceived stress.
PSS-10 Score at Post-Intervention | Month 2
  The PSS-10 is used to measure perceived stress over the past month. Items are rated on a 5-point scale ranging from 0 (never) to 4 (very often). Total scores range from 0-40; higher scores indicate greater levels of perceived stress.
PSS-10 Score at Follow-Up | Month 6
  The PSS-10 is used to measure perceived stress over the past month. Items are rated on a 5-point scale ranging from 0 (never) to 4 (very often). Total scores range from 0-40; higher scores indicate greater levels of perceived stress.
PHQ-9 Score at Baseline | Baseline
  The PHQ-9 assesses depressive symptoms in the past two weeks. Each of the nine items is rated on a four-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.
PHQ-9 Score at Post-Intervention | Month 2
  The PHQ-9 assesses depressive symptoms in the past two weeks. Each of the nine items is rated on a four-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.
PHQ-9 Score at Follow-Up | Month 6
  The PHQ-9 assesses depressive symptoms in the past two weeks. Each of the nine items is rated on a four-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-27 with recommended cutoffs for mild (5-9), moderate (10-14), moderately severe (15-19) and severe (≥20) depressive symptoms. A PHQ-9 score of <5 indicates absence of clinically significant depressive symptoms.
GAD-7 Score at Baseline | Baseline
  The GAD-7 measures anxiety symptoms in the past 2 weeks. Each item is rated on a four-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with recommended cutoffs for mild (5-9), moderate (10-14), and severe (15-21) anxiety. A score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder.
GAD-7 Score at Post-Intervention | Month 2
  The GAD-7 measures anxiety symptoms in the past 2 weeks. Each item is rated on a four-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with recommended cutoffs for mild (5-9), moderate (10-14), and severe (15-21) anxiety. A score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder.
GAD-7 Score at Follow-Up | Month 6
  The GAD-7 measures anxiety symptoms in the past 2 weeks. Each item is rated on a four-point scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0-21 with recommended cutoffs for mild (5-9), moderate (10-14), and severe (15-21) anxiety. A score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder.
Sleep-Quality Score at Baseline | Baseline
  Participants will rate their sleep quality over the previous 1-week period using a 5-point Likert scale, where 1 = very poor, 2 = poor, 3 = fair, 4 = good, and 5 = very good.
Sleep-Quality Score at Post-Intervention | Month 2
  Participants will rate their sleep quality over the previous 1-week period using a 5-point Likert scale, where 1 = very poor, 2 = poor, 3 = fair, 4 = good, and 5 = very good.
Sleep-Quality Score at Follow-Up | Month 6
  Participants will rate their sleep quality over the previous 1-week period using a 5-point Likert scale, where 1 = very poor, 2 = poor, 3 = fair, 4 = good, and 5 = very good.
Average Sleep Duration at Baseline | Baseline
  Participants will complete 1 week of sleep assessments to track the amount of sleep per night. A FitBit watch will also be used to help track sleep duration.
Average Sleep Duration at Post-Intervention | Month 2
  Participants will complete 1 week of sleep assessments to track the amount of sleep per night. A FitBit watch will also be used to help track sleep duration.
Average Sleep Duration at Follow-Up | Month 6
  Participants will complete 1 week of sleep assessments to track the amount of sleep per night. A FitBit watch will also be used to help track sleep duration.
Patient Reported Outcomes Measurement Information System (PROMIS-10) Score at Baseline | Baseline
  PROMIS-10 measures physical, mental, and social functioning health. The raw score is the sum of responses and is converted to a T-score ranging from 0-100 with an average score of 50. Higher scores indicate greater overall health.
PROMIS-10 Score at Post-Intervention | Month 2
  PROMIS-10 measures physical, mental, and social functioning health. The raw score is the sum of responses and is converted to a T-score ranging from 0-100 with an average score of 50. Higher scores indicate greater overall health.
PROMIS-10 Score at Follow-Up | Month 6
  PROMIS-10 measures physical, mental, and social functioning health. The raw score is the sum of responses and is converted to a T-score ranging from 0-100 with an average score of 50. Higher scores indicate greater overall health.
Seattle Angina Questionnaire (SAQ-7) Score at Baseline | Baseline
  The 7-item SAQ measures disease-specific health over the prior four weeks in patients with coronary artery disease (CAD). The SAQ-7 produces a summary score ranging from 0-100, where higher scores indicate better disease specific health status.
SAQ-7 Score at Post-Intervention | Month 2
  The 7-item SAQ measures disease-specific health over the prior four weeks in patients with CAD. The SAQ-7 produces a summary score ranging from 0-100, where higher scores indicate better disease specific health status.
SAQ-7 Score at Follow-Up | Month 6
  The 7-item SAQ measures disease-specific health over the prior four weeks in patients with CAD. The SAQ-7 produces a summary score ranging from 0-100, where higher scores indicate better disease specific health status.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Tanya.Spruill@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Tanya.Spruill@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.